CLINICAL TRIAL: NCT02478606
Title: Comparison of Four Weeks of Passive Static Stretching and Proprioceptive Neuromuscular Facilitation (PNF) in Musculoskeletal Aspects of the Hamstrings: a Randomized Controlled Trial
Brief Title: Passive Static Stretching and Proprioceptive Neuromuscular Facilitation in Musculoskeletal Aspects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Anelize Cini, Student of post graduate, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1.102.297
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-06

CONDITIONS: Flexibility; Range of Motion
Keywords: Lower Extremity; Muscle Stretching Exercises; Muscle Strength; Static Stretching; Proprioceptive Neuromuscular Facilitation (PNF) Stretching; Muscle Strength Dynamometer
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Control Group (No Intervention): Without intervention
- Static Group (Experimental): Will receive passive static stretching in hamstring muscle
  Interventions: Other: Muscle Stretching Exercises
- PNF Group (Experimental): Will receive passive proprioceptive neuromuscular facilitation stretching in hamstring muscle
  Interventions: Other: Muscle Stretching Exercises

INTERVENTIONS:
Other: Muscle Stretching Exercises — The training consists of a four-week program of passive stretching exercise with three times week/sessions with interval of 48 hours between them. Each session will consist of carrying out a single repetition of stretching exercise with 30s of duration, static or PNF, according to the group to which voluntary membership. The two lower members receive training but only the lower limb data drawn will be used for analysis.
  Other Names: Passive Static Stretching; Proprioceptive neuromuscular facilitation
  Arms: PNF Group; Static Group

SUMMARY:
This study investigates the influence of two different stretching techniques on the flexibility of the muscles that are in the posterior thigh, after a training period.

The study will last for six weeks where the volunteers need to go to the lab twice for evaluation, and for four weeks, three times a week for the application of stretching training.

Evaluation before and after the training period consists of applying hip and knee flexibility tests, evaluation of strength, muscle activation and muscle architecture. The Flexibility tests are: (1) Straight Leg Raise Flexibility Test (SLR), where the volunteer will be positioned supine on a stretcher. Then the appraiser will perform hip flexion keeping the knee extended and relaxed foot to the angle at which the person refer discomfort while the contralateral limb remain firmly leaning on the table; (2) Modified Passive knee extension (TEJ), where the volunteer will be positioned supine on a stretcher. The assessor shall determine the hip member to be rated at 90º and perform knee extension to the angle at which the person refer discomfort. The contralateral limb remain firmly leaning on the table.

For the evaluation of muscle strength the volunteer had sat on equipment, makes five repetitions of bending and straightening the knee to familiarize yourself with the equipment and after will make other five replicates doing maximum strength.

To evaluate the electrical activity will be the depilation of the skin with a razor and cleaning with an alcohol swab after adhesive electrodes will be placed for collection of muscle activity, the electrodes do not emit shocks.

The muscle architecture will be assessed via a ultrasound , to its use the use of a water soluble gel to improve the machine's skin contact is required.

For the intervention, the stretching will be held in both legs, where the volunteer will remain lying on a stretcher with fixed trunk with velcro straps and the researcher will carry out the elongation raising the leg drawn to the moment of discomfort the volunteer will refer and will remain for 30 seconds (s) in case he belongs to passive static stretching group, if the stretching group of proprioceptive neuromuscular facilitation, will be in the same position, but before the 30s of stretching, he you will have to push against during 6s to lower leg against the researcher.

If he belongs to the control group, have only two trips to the laboratory for testing, will make an initial assessment and after four weeks will return to perform the tests again, in the period between assessments will not need to go to the lab because it does not make intervention elongation.

It is possible that there discomfort during flexibility testing, strength testing and stretching training. After the tests can still experience muscle pain should disappear within 48 hours. The risks of research are minimal, not exceeding those of a strength training session and stretching.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Aged between 20 and 30 years;
* Be sedentary as classification of the International Physical Activity Questionnaire (IPAQ);
* Make Use of oral contraceptives;
* Body Mass Index range 18 to 24.

Exclusion Criteria:

* Provided history of musculoskeletal injury or surgery of the lower limbs;
* Provide continuous pain in the legs or lower back pain;
* Make use of painkillers, anti-inflammatory and / or muscle relaxant;
* Being in pregnancy;
* Present laxity ligament;
* Achieve zero degrees of extension in Knee Extension Test Modified.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change of Range of motion | Participants will be followed for the duration of stretching training, an average of six weeks
  Flexibility of the hamstring muscles is defined as the range of motion achieved in the Straight Leg Raising Test and modified Knee Extension Test

SECONDARY OUTCOMES:
Change of Force hamstring | Participants will be followed for the duration of stretching training, an average of six weeks
  Will be referred to as the peak torque (N.m.) isometric, concentric and eccentric isokinetic assessment with a dynamometer isokinetic.
Change of Muscle electrical activation | Participants will be followed for the duration of stretching training, an average of six weeks
  Is defined as the value Root Mean Square (RMS) of the vastus lateralis, rectus femoris and biceps femoris obtained during the tests of muscular strength and flexibility through a Electromyograph.
Change of Muscle Architecture | Participants will be followed for the duration of stretching training, an average of six weeks
  Will be represented through the issue of length and muscle thickness measured by ultrasound.